CLINICAL TRIAL: NCT04247074
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of QM1114-DP for the Treatment of Moderate to Severe Lateral Canthal Lines and Glabellar Lines Alone or in Combination
Brief Title: Treatment of Moderate to Severe Lateral Canthal Lines and Glabellar Lines Alone or in Combination
Acronym: READY-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 43QM1902
Record Dates: First submitted 2020-01-07; First posted 2020-01-29 (Actual); Results first posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-06

CONDITIONS: Glabellar Frown Lines (GL); Lateral Canthal Lines (LCL)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- QM1114-DP in the LCL + Placebo in the GL (Experimental): QM1114-DP, a Botulinum Toxin Type A (BoNT-A) ; Mode of administration: intramuscular injection
  Interventions: Biological: botulinum toxin neuromodulator; Biological: Placebo
- Placebo in the LCL and GL (Placebo Comparator): A buffered solution; Mode of administration:
  intramuscular injection
  Interventions: Biological: Placebo
- Placebo in the LCL + QM1114-DP in the GL (Experimental): QM1114-DP, a Botulinum Toxin Type A (BoNT-A) or placebo Mode of administration: intramuscular injection
  Interventions: Biological: botulinum toxin neuromodulator; Biological: Placebo
- QM1114-DP in the LCL + GL (Experimental): QM1114-DP, a Botulinum Toxin Type A (BoNT-A) ; Mode of administration: intramuscular injection
  Interventions: Biological: botulinum toxin neuromodulator

INTERVENTIONS:
Biological: botulinum toxin neuromodulator — QM1114-DP will be injected into either the LCL, GL, or both the LCL and GL
  Other Names: QM1114-DP
  Arms: Placebo in the LCL + QM1114-DP in the GL; QM1114-DP in the LCL + GL; QM1114-DP in the LCL + Placebo in the GL
Biological: Placebo — Placebo will be injected into either the LCL, GL, or both the LCL and GL
  Arms: Placebo in the LCL + QM1114-DP in the GL; Placebo in the LCL and GL; QM1114-DP in the LCL + Placebo in the GL

SUMMARY:
This study is designed to evaluate the safety and efficacy of a single dose of QM1114-DP for the treatment of moderate to severe LCL and moderate to severe GL, alone or in combination.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older.
2. Moderate to severe LCL at maximum smile as assessed by the Investigator.
3. Moderate to severe LCL at maximum smile as assessed by the subject.
4. Moderate to severe GL at maximum frown as assessed by the Investigator.
5. Moderate to severe GL at maximum frown as assessed by the subject

Exclusion Criteria:

1. Previous use of any Botulinum toxin in facial areas within 9 months prior to study treatment.
2. Female who is pregnant, breast feeding, or intends to conceive a child during the study.
3. Known allergy or hypersensitivity to any component of the investigational product (QM1114-DP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - Clinical Testing of Beverly Hills, Encino, California
  - Ava MD, Santa Monica, California
  - Skin Care & Laser Physicians of Beverly Hills, West Hollywood, California
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - Baumann Cosmetic & Research Institute, Inc, Miami, Florida
  - Washington Institute of Dermatologic Laser Surgery, Chevy Chase, Maryland
  - Maryland Dermatology, Laser, Skin & Vein Institute, Hunt Valley, Maryland
  - Skin Specialists, PC, Omaha, Nebraska
  - Lorenc Aesthetic Plastic Surgery Center, New York, New York
  - Elite Aesthetic Research, Cincinnati, Ohio
  - The Westlake Dermatology Clinical Research, Austin, Texas
- Bertucci Medspa, Inc, Woodbridge, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- QM1114-DP in the LCL + Placebo in the GL: QM1114-DP, a Botulinum Toxin Type A (BoNT-A) or placebo. Mode of administration: intramuscular injection Botulinum toxin neuromodulator, QM1114-DP, will be injected into the LCL. Placebo, a buffered solution, will be injected the GL.
  QM1114-DP LCL dosage:
  60 units, 0.6 mL total, 0.1 mL per LCL injection point
  Placebo GL dosage:
  0.5 mL total, 0.1 mL per GL injection point
- Placebo in the LCL and GL: Placebo, a buffered solution. Mode of administration: intramuscular injection. Placebo will be injected into both the LCL and GL.
  Placebo LCL dosage:
  0.6 mL total, 0.1 mL per LCL injection point
  Placebo GL dosage:
  0.5 mL total, 0.1 mL per GL injection point
- Placebo in the LCL + QM1114-DP in the GL: QM1114-DP, a Botulinum Toxin Type A (BoNT-A) or placebo. Mode of administration: intramuscular injection. Placebo, a buffered solution, will be injected into the LCL. Botulinum toxin neuromodulator, QM1114-DP, will be injected into the GL.
  Placebo LCL dosage:
  0.6 mL total, 0.1 mL per LCL injection point
  QM1114-DP GL dosage:
  50 units, 0.5 mL total, 0.1 mL per GL injection point
- QM1114-DP in the LCL + GL: QM1114-DP, a Botulinum Toxin Type A (BoNT-A). Mode of administration: intramuscular injection. Botulinum toxin neuromodulator: QM1114-DP will be injected into both the LCL and GL.
  QM1114-DP LCL dosage:
  60 units, 0.6 mL total, 0.1 mL per LCL injection point
  QM1114-DP GL dosage:
  50 units, 0.5 mL total, 0.1 mL per GL injection point
Period: Overall Study
Arm/Group | QM1114-DP in the LCL + Placebo in the GL | Placebo in the LCL and GL | Placebo in the LCL + QM1114-DP in the GL | QM1114-DP in the LCL + GL
Started | 126 | 59 | 113 | 115
Completed | 121 | 52 | 106 | 107
Not Completed | 5 | 7 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- QM1114-DP in the LCL + Placebo in the GL: QM1114-DP, a Botulinum Toxin Type A (BoNT-A) or placebo. Mode of administration: intramuscular injection. Botulinum toxin neuromodulator, QM1114-DP, will be injected into the LCL. Placebo, a buffered solution, will be injected the GL.
  QM1114-DP LCL dosage:
  60 units, 0.6 mL total, 0.1 mL per LCL injection point
  Placebo GL dosage:
  0.5 mL total, 0.1 mL per GL injection point
- Total: Total of all reporting groups
Arm/Group | QM1114-DP in the LCL + Placebo in the GL | Placebo in the LCL and GL | Placebo in the LCL + QM1114-DP in the GL | QM1114-DP in the LCL + GL | Total
Number analyzed (Participants) | 126 | 59 | 113 | 115 | 413
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (10.44) | 49.8 (50.0) | 50.4 (9.77) | 50.5 (10.63) | 50.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We had one subject randomized to Placebo/Placebo group but they weren't treated (Subject was randomized in error and discontinued prior to receiving treatment.). Therefore, they are not included in the ITT or Safety populations.
  Participants
    number analyzed (Participants) | 126 | 58 | 113 | 115 | 412
    Female | 113 | 55 | 103 | 97 | 368
    Male | 13 | 3 | 10 | 18 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: We had one subject randomized to Placebo/Placebo group but they weren't treated (Subject was randomized in error and discontinued prior to receiving treatment.). Therefore, they are not included in the ITT or Safety populations.
  Participants
    number analyzed (Participants) | 126 | 58 | 113 | 115 | 412
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 1 | 0 | 1 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
    Black or African American | 6 | 2 | 7 | 6 | 21
    White | 115 | 54 | 105 | 105 | 379
    More than one race | 1 | 0 | 0 | 2 | 3
    Unknown or Not Reported | 3 | 1 | 0 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a ≥ 2-grade Improvement From Baseline on the Glabellar Lines Investigator and Subject Assessments at Maximum Frown
Description: Investigator 4-point Photographic Scale of Glabellar Line Severity represents the severity of GL from none (grade 0), mild (grade 1), moderate (grade 2) to severe (grade 3). Each grade is depicted by an individual photograph and a descriptive text. The Investigators used the 4-point Photographic Scale for direct, live comparison with the subject's face at maximum frown.
  Subjects made their assessment of glabellar line severity independently of the Investigator's assessment. Subjects were asked to evaluate their GL at maximum frown by grading the GL severity from none (grade 0, smooth skin), mild (grade 1, fairly smooth skin), moderate (grade 2, frown lines) to severe (grade 3, deep frown lines).
Time Frame: Month 1
Population: Modified ITT population as actually randomized: All subjects ITT population who had an on-site Month 1 endpoint assessment conducted. The primary endpoint includes both LCL and GL analyses. The primary endpoint for GL success is dependent on results from 3 out of the 4 arms, which is provided. QM1114-DP in the LCL + Placebo analyses are presented in the next section as it is only relevant for the LCL endpoint success.
Measure: Count of Participants; unit: Participants
Groups:
- QM1114-DP in the LCL + GL (GL Data): QM1114-DP, a Botulinum Toxin Type A (BoNT-A). Mode of administration: intramuscular injection. Botulinum toxin neuromodulator: QM1114-DP will be injected into both the LCL and GL.
  QM1114-DP LCL dosage:
  60 units, 0.6 mL total, 0.1 mL per LCL injection point
  QM1114-DP GL dosage:
  50 units, 0.5 mL total, 0.1 mL per GL injection point
Arm/Group | Placebo in the LCL and GL | Placebo in the LCL + QM1114-DP in the GL | QM1114-DP in the LCL + GL (GL Data)
Number analyzed (Participants) | 55 | 106 | 108
Participants | 0 | 75 | 78
Statistical Analysis 1: Comparison: Placebo in the LCL and GL vs Placebo in the LCL + QM1114-DP in the GL vs QM1114-DP in the LCL + GL (GL Data); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

2. Primary Outcome: Percentage of Subjects With a ≥ 2-grade Improvement From Baseline on the Lateral Canthal Lines Investigator and Subject Assessments at Maximum Smile
Description: Investigator 4-point Photographic Scale of Lateral Canthal Line represents LCL severities from none (grade 0), mild (grade 1), moderate (grade 2), to severe (grade 3). Each grade is also depicted by an individual photograph and descriptive text. The Investigators used the LCL-ILA for direct, live comparison with the subject's face for grading LCL severity. Left and right LCL were assessed at maximum smile.
  Subject 4-point Photographic Scale of Lateral Canthal Line Severity represents LCL severities from Level 0, Level 1, Level 2, to Level 3. Each grade is also depicted by an individual photograph and descriptive text. Subjects made their assessments independently of the Investigator's assessment. Subjects evaluated their LCL severity (left and right side separately) at maximum smile.
Time Frame: Month 1
Population: Modified intent-to-treat population as actually randomized: All subjects in intent-to-treat population who had an on-site Month 1 primary endpoint assessment conducted.
Measure: Count of Participants; unit: Participants
Groups:
- QM1114-DP in the LCL + Placebo in the GL: QM1114-DP, a Botulinum Toxin Type A (BoNT-A) or placebo. Mode of administration: intramuscular injection. Botulinum toxin neuromodulator, QM1114-DP, will be injected into the LCL. Placebo, a buffered solution, will be injected the GL.
  QM1114-DP LCL dosage:
  60 units, 0.6 mL total, 0.1 mL per LCL injection point
  Placebo GL dosage:
  0.5 mL, total 0.1 mL per GL injection point
- QM1114-DP in the LCL + GL (LCL Data): QM1114-DP, a Botulinum Toxin Type A (BoNT-A). Mode of administration: intramuscular injection. Botulinum toxin neuromodulator: QM1114-DP will be injected into both the LCL and GL.
  QM1114-DP LCL dosage:
  60 units, 0.6 mL total, 0.1 mL per LCL injection point
  QM1114-DP GL dosage:
  50 units, 0.5 mL total, 0.1 mL per GL injection point
Arm/Group | QM1114-DP in the LCL + Placebo in the GL | Placebo in the LCL and GL | QM1114-DP in the LCL + GL (LCL Data)
Number analyzed (Participants) | 117 | 55 | 108
Participants | 53 | 0 | 59
Statistical Analysis 1: Comparison: QM1114-DP in the LCL + Placebo in the GL vs Placebo in the LCL and GL vs QM1114-DP in the LCL + GL (LCL Data); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Subjects With a 0 or 1 on the Glabellar Lines Investigator Scale at Maximum Frown
Time Frame: Month 1
Population: Intent to treat population (all subjects randomized and administered study product) as actually randomized, excluding remote assessments.
  The secondary endpoint includes both LCL and GL analyses. QM1114-DP in the LCL + Placebo in the GL group analyses are presented in the next section. This is also applicable for the combination treatment (QM1114-DP in the LCL + GL) LCL outcome results.
Measure: Count of Participants; unit: Participants
Groups:
- QM1114-DP in the LCL + GL: Botulinum Toxin Type A (BoNT-A). Mode of administration: intramuscular injection. Botulinum toxin neuromodulator: QM1114-DP will be injected into both the LCL and GL.
  QM1114-DP LCL dosage:
  60 units, 0.6 mL total, 0.1 mL per LCL injection point
  QM1114-DP GL dosage:
  50 units, 0.5 mL total, 0.1 mL per GL injection point
Arm/Group | Placebo in the LCL and GL | Placebo in the LCL + QM1114-DP in the GL | QM1114-DP in the LCL + GL
Number analyzed (Participants) | 51 | 103 | 106
Participants | 1 | 97 | 102
Statistical Analysis 1: Comparison: Placebo in the LCL and GL vs Placebo in the LCL + QM1114-DP in the GL vs QM1114-DP in the LCL + GL; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Percentage of Subjects Who Achieve Grade 0 or 1 in Lateral Canthal Line Investigator Scale at Maximum Smile.
Time Frame: Month 1
Population: Intent to treat population (all subjects randomized and administered study product) as actually randomized, excluding remote assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | QM1114-DP in the LCL + Placebo in the GL | Placebo in the LCL and GL | QM1114-DP in the LCL + GL (LCL Data)
Number analyzed (Participants) | 113 | 51 | 106
Participants | 89 | 10 | 89
Statistical Analysis 1: Comparison: QM1114-DP in the LCL + Placebo in the GL vs Placebo in the LCL and GL vs QM1114-DP in the LCL + GL (LCL Data); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 6 months
Description: 3 subjects had a randomization error which is why there is a difference in the Participant Flow (All Subjects Population) and the Adverse Events (Safety Population)
  Safety Population: All subjects who were administered the study product; subjects were analyzed according to as-treated principle.
Groups:
- QM1114-DP in the LCL + Placebo in the GL: AEs are not collected separately for each type of treatment in each arm.
  QM1114-DP, a Botulinum Toxin Type A (BoNT-A) or placebo. Mode of administration: intramuscular injection.
  Botulinum toxin neuromodulator, QM1114-DP, will be injected into the LCL. Placebo, a buffered solution, will be injected the GL.
  QM1114-DP LCL dosage:
  60 units, 0.6 mL total, 0.1 mL per LCL injection point
  Placebo GL dosage:
  0.5 mL total, 0.1 mL per GL injection point
- Placebo in the LCL and GL: AEs are not collected separately for each type of treatment in each arm.
  Placebo, a buffered solution. Mode of administration: intramuscular injection. Placebo will be injected into both the LCL and GL.
  Placebo LCL dosage:
  0.6 mL total, 0.1 mL per LCL injection point
  Placebo GL dosage:
  0.5 mL total, 0.1 mL per GL injection point
- Placebo in the LCL + QM1114-DP in the GL: AEs are not collected separately for each type of treatment in each arm.
  QM1114-DP, a Botulinum Toxin Type A (BoNT-A) or placebo. Mode of administration: intramuscular injection. Placebo, a buffered solution, will be injected into the LCL.
  Botulinum toxin neuromodulator, QM1114-DP, will be injected into the GL.
  Placebo LCL dosage:
  0.6 mL total, 0.1 mL per LCL injection point
  QM1114-DP GL dosage:
  50 units, 0.5 mL total, 0.1 mL per GL injection point
- QM1114-DP in the LCL + GL: AEs are not collected separately for each type of treatment in each arm.
  QM1114-DP, a Botulinum Toxin Type A (BoNT-A). Mode of administration: intramuscular injection. Botulinum toxin neuromodulator: QM1114-DP will be injected into both the LCL and GL.
  QM1114-DP LCL dosage:
  60 units, 0.6 mL total 0.1 mL per LCL injection point
  QM1114-DP GL dosage:
  50 units, 0.5 mL total, 0.1 mL per GL injection point
Arm/Group | QM1114-DP in the LCL + Placebo in the GL | Placebo in the LCL and GL | Placebo in the LCL + QM1114-DP in the GL | QM1114-DP in the LCL + GL
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/58 | 0/116 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/123 | 1/58 | 1/116 | 1/115
Other Adverse Events (participants affected / at risk) | 9/123 | 6/58 | 18/116 | 9/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QM1114-DP in the LCL + Placebo in the GL (N=123) | Placebo in the LCL and GL (N=58) | Placebo in the LCL + QM1114-DP in the GL (N=116) | QM1114-DP in the LCL + GL (N=115)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QM1114-DP in the LCL + Placebo in the GL (N=123) | Placebo in the LCL and GL (N=58) | Placebo in the LCL + QM1114-DP in the GL (N=116) | QM1114-DP in the LCL + GL (N=115)
COVID-19 (Infections and infestations) | 4 (4) | 4 (4) | 6 (6) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 6 (6) | 4 (4)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Injection site bruising (General disorders) | 2 (2) | 1 (2) | 3 (3) | 2 (2)
Injection site pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT04247074/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT04247074/SAP_001.pdf